CLINICAL TRIAL: NCT00973596
Title: Swiss Venous Thromboembolism Cohort Study of Elderly Patients With Acute Venous Thromboembolism
Brief Title: The Swiss Venous Thromboembolism Cohort 65+
Acronym: SWITCO65+
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Drahomir Aujesky, Director of the Division of General Internal Medicine, University of Bern
Other Study IDs: 33CSCO-122 659/139 470
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective multicenter cohort study is to examine long-term medical outcomes, quality of life, and medical resource utilization in elderly patients (>= 65 years) with acute venous thromboembolism (i.e., acute pulmonary embolism and/or deep vein thrombosis)

ELIGIBILITY:
Inclusion Criteria:

* Objectively confirmed acute pulmonary embolism and/or deep vein thrombosis
* Age >=65 years

Exclusion Criteria:

* Thrombosis at a different site than lower limb
* Catheter-related thrombosis
* Insufficient spoken language ability in German or French
* Follow-up not possible (e.g., terminally ill patients)
* Informed consent not possible (e.g., severe dementia)
* Prior enrolment in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Outpatients and inpatients with acute venous thromboembolism from 9 Swiss university and non-university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism recurrence | 3-48 months

SECONDARY OUTCOMES:
Overall mortality | 3-48 months
Major bleeding | 3-48 months
Post-thrombotic syndrome | 3-48 months
Generic and disease-specific health-related quality of life | 3-48 months
Medical resource utilization | 3-48 months

CONTACTS AND LOCATIONS:
Locations (9):
- Switzerland (9):
  - Kantonsspital Baden, Baden
  - University Hospital of Basel, Basel
  - University Hospital of Bern, Bern
  - Kantonsspital Frauenfeld, Frauenfeld
  - University Hospital of Geneva, Geneva
  - University Hospital of Lausanne, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital of Zurich, Zurich

REFERENCES:
- [Derived] Jaquet E, Tritschler T, Stalder O, Limacher A, Mean M, Rodondi N, Aujesky D. Prediction of short-term prognosis in elderly patients with acute pulmonary embolism: validation of the RIETE score. J Thromb Haemost. 2018 Jul;16(7):1313-1320. doi: 10.1111/jth.14137. Epub 2018 May 30. PMID 29733493
- [Derived] Lauber S, Limacher A, Tritschler T, Stalder O, Mean M, Righini M, Aschwanden M, Beer JH, Frauchiger B, Osterwalder J, Kucher N, Lammle B, Cornuz J, Angelillo-Scherrer A, Matter CM, Husmann M, Banyai M, Staub D, Mazzolai L, Hugli O, Rodondi N, Aujesky D. Predictors and Outcomes of Recurrent Venous Thromboembolism in Elderly Patients. Am J Med. 2018 Jun;131(6):703.e7-703.e16. doi: 10.1016/j.amjmed.2017.12.015. Epub 2018 Jan 4. PMID 29307536
- [Derived] Seiler E, Limacher A, Mean M, Beer HJ, Osterwalder J, Frauchiger B, Righini M, Aschwanden M, Matter CM, Banyai M, Kucher N, Staub D, Lammle B, Rodondi N, Squizzato A, Aujesky D. Derivation and validation of a novel bleeding risk score for elderly patients with venous thromboembolism on extended anticoagulation. Thromb Haemost. 2017 Aug 24;117(10). doi: 10.1160/TH17-03-0162. Online ahead of print. PMID 28837210
- [Derived] Hofmann E, Limacher A, Mean M, Kucher N, Righini M, Frauchiger B, Beer JH, Osterwalder J, Aschwanden M, Matter CM, Banyai M, Egloff M, Hugli O, Staub D, Bounameaux H, Rodondi N, Aujesky D. Echocardiography does not predict mortality in hemodynamically stable elderly patients with acute pulmonary embolism. Thromb Res. 2016 Sep;145:67-71. doi: 10.1016/j.thromres.2016.07.014. Epub 2016 Jul 27. PMID 27498122
- [Derived] Vuilleumier N, Simona A, Mean M, Limacher A, Lescuyer P, Gerstel E, Bounameaux H, Aujesky D, Righini M. Comparison of Cardiac and Non-Cardiac Biomarkers for Risk Stratification in Elderly Patients with Non-Massive Pulmonary Embolism. PLoS One. 2016 May 24;11(5):e0155973. doi: 10.1371/journal.pone.0155973. eCollection 2016. PMID 27219621
- [Derived] Tritschler T, Mean M, Limacher A, Rodondi N, Aujesky D. Predicting recurrence after unprovoked venous thromboembolism: prospective validation of the updated Vienna Prediction Model. Blood. 2015 Oct 15;126(16):1949-51. doi: 10.1182/blood-2015-04-641225. Epub 2015 Sep 4. PMID 26341256
- [Derived] Frey PM, Mean M, Limacher A, Jaeger K, Beer HJ, Frauchiger B, Aschwanden M, Rodondi N, Righini M, Egloff M, Osterwalder J, Kucher N, Angelillo-Scherrer A, Husmann M, Banyai M, Matter CM, Aujesky D. Physical activity and risk of bleeding in elderly patients taking anticoagulants. J Thromb Haemost. 2015 Feb;13(2):197-205. doi: 10.1111/jth.12793. Epub 2014 Dec 30. PMID 25403550